CLINICAL TRIAL: NCT01936935
Title: A Randomized, Controlled, Crossover Trial to Assess the Effects of Dairy Intake on Insulin Sensitivity and β-Cell Function in Men and Women at Risk for Diabetes Who Are Habitual Consumers of High Sugar Beverages
Brief Title: Clinical Trial to Assess the Effects of Dairy on Insulin Sensitivity and β-Cell Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Provident Clinical Research (Other)
Collaborators: BioFortis (Other); Dairy Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: PRV-1222
Record Dates: First submitted 2013-09-03; First posted 2013-09-06 (Estimated); Last update posted 2023-12-04 (Actual); Status verified 2013-09

CONDITIONS: Diabetes
Keywords: Insulin sensitivity
MeSH Terms: conditions — Diabetes Mellitus; Insulin Resistance | interventions — Sugar-Sweetened Beverages

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low-fat dairy (Experimental): 3 servings/d of low-fat dairy
  Interventions: Other: Low-fat dairy
- Sugar-sweetened beverages (Placebo Comparator): 3 servings/d of sugar-sweetened foods
  Interventions: Other: Sugar-sweetened beverages

INTERVENTIONS:
Other: Low-fat dairy — 2 servings/d of 2% non-flavored, unsweetened milk + 1 serving/d sweetened low-fat yogurt
  Arms: Low-fat dairy
Other: Sugar-sweetened beverages — 2 servings/d of non-diet soda + 1 serving/d of non-dairy pudding
  Arms: Sugar-sweetened beverages

SUMMARY:
The aim of this trial is to evaluate the effects of dairy product consumption on insulin sensitivity and pancreatic β-cell function in men and women at risk for the development of type 2 diabetes mellitus (T2DM) who habitually consume beverages high in sugar (non-diet sodas and fruit juice cocktails).

ELIGIBILITY:
Inclusion Criteria:

* subject is male or female, 18-74 yrs of age, inclusive
* subject reports habitual consumption of ≥2 servings/d of high-sugar beverages (e.g., non-diet soda, fruit juice cocktails)
* subject has waist circumference ≥33.0 inches for women and ≥36.0 inches for men
* subject is at risk for development of type 2 diabetes mellitus (T2DM), based on 1 or more of the following: fasting glucose 100-125 mg/dL; glycosylated hemoglobin 5.7-6.4%, or ≥20% risk of developing diabetes in the next 7.5 yrs based on the San Antonio Heart Study prediction equation
* subject has a score of 7-10 on the Vein Access Scale at screening
* subject is normally active and judged to be in good health on the basis of medical history, physical examination and routine lab tests
* if female, subject is willing to schedule treatment visits during the follicular phase of the menstrual cycle, defined as days 1-14, where day 1 is 1st day of menses
* subject has a menstrual cycle duration ranging in length form 24-36 d (if premenopausal)
* subject is willing to maintain a stable body weight and follow his/her habitual diet and exercise pattern, except for inclusion of study product, throughout the trial
* subject is willing to maintain his or her habitual intake of coffee, tea, and alcoholic beverages throughout the trial
* subject agrees to limit intake of non-study related dairy products to ≤1 serving per day during each treatment period
* subject is ambulatory and willing to refrain from vigorous physical activity and consumption of alcoholic beverages 24 h prior to each test day
* subject has no plans to change smoking habits during the study period
* subject is willing to abstain from tobacco use 1 h prior to and during visits on LMTT test days
* subject has no health conditions that would prevent him/her from fulfilling the study requirements as judged by the Investigator on the basis of medical history and routine lab test results

Exclusion Criteria:

* subject has abnormal lab test results of clinical importance, including, but not limited to, TG ≥400 mg/dL, fasting creatinine ≥1.5 mg/dL, alanine aminotransferase or aspartate aminotransferase ≥1.5 times the upper limit of normal at screening
* subject has a body mass index ≥45.0 kg/m2
* subject has fasting blood glucose ≥126 mg/dL at screening or known diabetes mellitus (type 1 or T2DM)
* subject has a habitual intake of ≥4 servings/d of dairy food and beverages
* subject has known allergy or sensitivity to study product or any ingredients of study product. Subjects with lactose intolerance will be allowed to use products such as Lactaid dietary supplements
* subject has a history of coronary heart disease, congestive heart failure, or serious ventricular dysrhythmias (ventricular tachycardia or fibrillation)
* subject has a change in body weight of >4.5 kg within 4 weeks of screening
* subject uses medications known to influence carbohydrate metabolism
* subject has recent use of antibiotics
* subject has an active infection
* subject has unstable use of anti-hypertensive medications, thyroid hormone replacement, or lipid-altering drugs within 4 weeks of screening
* subject has unstable use of lipid-altering foods or dietary supplements within 4 weeks of screening
* subject uses niacin at doses >200 mg/d within 4 weeks of screening
* subject has history of extreme dietary habits, e.g., Atkins, high protein
* subject has a history or presence of clinically important endocrine, cardiac, renal, hepatic, pulmonary, biliary, pancreatic, gastrointestinal, or neurologic disorders that could interfere with interpretation of study results
* subject has history of dysphagia, swallowing disorders, or intestinal motility disorders
* subject has history of cancer
* subject has uncontrolled hypertension at screening (systolic blood pressure ≥160 mm Hg or diastolic blood pressure ≥100 mm Hg)

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2012-09 (Actual); Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Matsuda Insulin Sensitivity Index (MISI) | 6 weeks
  MISI calculated from glucose and insulin data obtained during a liquid meal tolerance test (LMTT). MISI = 10,000 divided by the square root of the quantity of fasting glucose x fasting insulin x mean post-load glucose from samples collected at 30, 60, 90 and 120 min after the start of the liquid meal x mean post-load insulin from samples collected at 30, 60, 90 and 120 min after the start of the liquid meal

SECONDARY OUTCOMES:
Waist circumference | 6 weeks
  Measured using a non-stretch anthropometric tape
Blood pressure | 6 weeks
  Standardized vital signs measurements will include resting blood pressure and pulse measured using an automated blood pressure measurement device.
Fasting and 2-hr LMTT insulin and glucose concentrations | 6 weeks
  During the LMTT subjects consume a liquid meal load (two-8 oz servings of Ensure®, Ross Products Division, Abbott Laboratories, Columbus, Ohio), and blood samples will be obtained at t = -10, 30, 60, 90, and 120 min ± 5 min where t = 0 min is the start of meal consumption. Serum insulin and plasma glucose concentrations will be measured in fasting (-10 min) and 2 hr (120 min) samples.
Homeostasis model assessment of insulin resistance (HOMA-IR) | 6 weeks
  HOMA-IR = the quantity of fasting glucose in mg/dL x fasting insulin in microunits/mL divided by 405
Homeostasis model assessment of beta-cell function (HOMA%B) | 6 weeks
  HOMA%B = 360 x fasting insulin in microunits/mL divided by fasting glucose in mg/dL minus 63
Glucose total area under the curve (AUC) from 0-120 min | 6 weeks
  Glucose total AUC 0-120 min will be calculated using the trapezoidal rule on glucose concentrations in blood samples collected at -10, 30, 60, 90, and 120 min where 0 min is the start of the liquid meal consumption in the LMTT.
Insulin total AUC 0-120 min | 6 weeks
  Insulin total AUC 0-120 min will be calculated using the trapezoidal rule on insulin concentrations in blood samples collected at -10, 30, 60, 90, and 120 min where 0 min is the start of the liquid meal consumption in the LMTT.
30 min Δ insulin/Δ glucose | 6 weeks
  Change in insulin from baseline to 30 min of the LMTT will be divided by the change in glucose from baseline to 30 min of the LMTT
AUC insulin/AUC glucose | 6 weeks
  AUC for insulin divided by the AUC for glucose
Disposition Index | 6 weeks
  Disposition index = MISI x the quantity of AUC for insulin divided by the AUC for glucose
Fasting plasma total cholesterol (total-C) | 6 weeks
Fasting plasma low-density lipoprotein cholesterol (LDL-C) | 6 weeks
  Calculated as LDL-C = total-C minus HDL-C minus the quantity of triglycerides (TG) divided by 5
Fasting plasma high-density lipoprotein cholesterol (HDL-C) | 6 weeks
Fasting plasma total-C/HDL-C | 6 weeks
  Calculated as total-C concentration divided by HDL-C concentration
Fasting plasma non-HDL-C | 6 weeks
  Calculated as non-HDL-C = total-C minus HDL-C
Fasting plasma TG | 6 weeks
Serum 25-hydroxy vitamin D [25(OH)D] | 6 weeks
Plasma high-sensitivity C-reactive protein (hs-CRP) | 6 weeks

OTHER OUTCOMES:
Mean circulating glucose level | 6 weeks
  Mean circulating glucose level will be measured over 24 h in the continuous glucose monitoring (CGM) subset of subjects
Mean daytime glucose values | 6 weeks
  Mean daytime glucose values (6 am to 8 pm) measured in the CGM subset of subjects
Mean evening/nighttime glucose values | 6 weeks
  Mean evening/nighttime glucose values (8 pm to 6 am) measured in the CGM subset of subjects
Mean peak postprandial glucose | 6 weeks
  Mean peak postprandial glucose values during CGM after the lunch and dinner meals

CONTACTS AND LOCATIONS:
Overall Officials: Kevin C Maki, PhD, Study Director — Biofortis Clinical Research, Inc.
Locations (1):
- Provident Clinical Research (now Biofortis), Addison, Illinois, United States

REFERENCES:
- [Derived] Maki KC, Nieman KM, Schild AL, Kaden VN, Lawless AL, Kelley KM, Rains TM. Sugar-sweetened product consumption alters glucose homeostasis compared with dairy product consumption in men and women at risk of type 2 diabetes mellitus. J Nutr. 2015 Mar;145(3):459-66. doi: 10.3945/jn.114.204503. Epub 2015 Jan 7. PMID 25733460